CLINICAL TRIAL: NCT04869735
Title: Impact of Information About Booster Vaccination Against DTPolio at 25 Years on This Booster Vaccination's Realization
Acronym: Info-Vac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-003-Info-Vac
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-04

CONDITIONS: Vaccination
Keywords: Booster vaccination; Adult; Information; DTPolio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With information about booster vaccination: Adults aged 25 years in 2020 without delivery of DTPolio vaccine in 2019 or 2020, to whom information concerning this vaccination is given
  Interventions: Other: Data collection: DTPolio vaccine delivery
- Without information about booster vaccination: Adults aged 25 years in 2020 without delivery of DTPolio vaccine in 2019 or 2020, to whom information concerning this vaccination is not given.
  Interventions: Other: Data collection: DTPolio vaccine delivery

INTERVENTIONS:
Other: Data collection: DTPolio vaccine delivery — "with information about booster vaccination" group: Sending of information concerning booster vaccination against DTPolio at 25 years using letters, emails and SMS "without information about booster vaccination" group: no intervention

SUMMARY:
The aim of vaccination is to protect the patient against disease by stimulating his immune system. DTPolio is a tetravalent vaccine providing protection against pertussis, diphtheria, tetanus and polio.

In France, the vaccination schedule sets the vaccination recommendations applicable to people according to their age. In this schedule, a booster of DTPolio at the age of 25 is recommended.

The vaccination coverage for patients over 16 years of age is insufficient in France.

DETAILED DESCRIPTION:
The aim of the study is to evaluate impact of information about booster vaccination against DTPolio at 25 years on this booster vaccination's realization.

ELIGIBILITY:
Inclusion Criteria:

* aged 25 years old in 2020
* without delivery of DTPolio vaccine in 2019 or 2020

Exclusion Criteria:

* None

Ages: 25 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People aged 25
Sampling Method: Non-Probability Sample
Enrollment: 2125 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
DTPolio vaccine delivery | 12 months
  DTPolio vaccine delivery by pharmacies within 12 months of sending information about booster vaccination against DTPolio at 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte VUILLEMIN, Principal Investigator — Université de Reims CHampahne-Ardenne
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France